CLINICAL TRIAL: NCT06252519
Title: Pharmacokinetic Profile of N-Acetyl Cysteine in Self-reported Healthy Men and Women
Brief Title: Pharmacokinetic Profile of N-Acetyl Cysteine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Nature Fusions (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PRO-FY2023-417
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Pharmacokinetics
Keywords: N-Acetyl Cysteine; N-Acetyl Cysteine Ethyl Ester

STUDY DESIGN:
Intervention Model Description: Randomized cross-over single-blinded study
Who Masked: Participant
Masking Description: Each treatment was assigned a letter and provided to subjects in a paper cup.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- NAC, then neuro-NAC, then Neuro-NAC XS (Experimental): Participants receive single dose of NAC while on controlled diet. One week later, participants receive 1 dose Neuro-NAC while on controlled diet. One week later, participants receive 1 dose Neuro-NAC XS while on controlled diet.
  Interventions: Dietary Supplement: NAC; Dietary Supplement: Neuro-NAC; Dietary Supplement: Neuro-NAC XS
- NAC, Neuro-NAC XS, then Neuro-NAC (Experimental): Participants receive single dose of NAC while on controlled diet. One week later, participants receive 1 dose Neuro-NAC XS while on controlled diet.
  One week later, participants receive 1 dose Neuro-NAC while on controlled diet.
  Interventions: Dietary Supplement: NAC; Dietary Supplement: Neuro-NAC; Dietary Supplement: Neuro-NAC XS
- Neuro-NAC, then NAC, then Neuro-NAC XS (Experimental): Participants receive single dose of Neuro-NAC while on controlled diet. One week later, participants receive 1 dose NAC while on controlled diet. One week later, participants receive 1 dose Neuro-NAC XS while on controlled diet.
  Interventions: Dietary Supplement: NAC; Dietary Supplement: Neuro-NAC; Dietary Supplement: Neuro-NAC XS
- Neuro-NAC, then Neuro-NAC XS, then NAC (Experimental): Participants receive single dose of Neuro-NAC while on controlled diet. One week later, participants receive 1 dose Neuro-NAC XS while on controlled diet.
  One week later, participants receive 1 dose NAC while on controlled diet.
  Interventions: Dietary Supplement: NAC; Dietary Supplement: Neuro-NAC; Dietary Supplement: Neuro-NAC XS
- Neuro-NAC XS, then NAC, then Neuro-NAC (Experimental): Participants receive single dose of Neuro-NAC XS while on controlled diet. One week later, participants receive 1 dose NAC while on controlled diet. One week later, participants receive 1 dose Neuro-NAC while on controlled diet.
  Interventions: Dietary Supplement: NAC; Dietary Supplement: Neuro-NAC; Dietary Supplement: Neuro-NAC XS
- Neuro-NAC XS, then Neuro-NAC, then NAC (Experimental): Participants receive single dose of Neuro-NAC XS while on controlled diet. One week later, participants receive 1 dose Neuro-NAC while on controlled diet. One week later, participants receive 1 dose NAC while on controlled diet.
  Interventions: Dietary Supplement: NAC; Dietary Supplement: Neuro-NAC; Dietary Supplement: Neuro-NAC XS

INTERVENTIONS:
Dietary Supplement: NAC — 1 375 mg capsule containing N-acetyl cysteine
Dietary Supplement: Neuro-NAC — 3 capsules containing a total of 375 mg N-Acetyl L-Cysteine Ethyl Ester
Dietary Supplement: Neuro-NAC XS — 3 capsules containing a total of 75 mcg Selenium, 150 mcg Molybdenum, 1800 mg Glycine, and 375 mg N-Acetyl L-Cysteine Ethyl Ester

SUMMARY:
The study compares three different formulations containing N-Acetyl Cysteine, with regards to acute absorption over a 24-hour period, following single ingestion. The formulations are traditional N-Acetyl Cysteine, N-Acetyl Cysteine Ethyl Ester, and a product containing a combination of N-Acetyl Cysteine Ethyl Ester, glycine, and two minerals with antioxidant potential (selenium and molybdenum) that might enhance the effect of N-Acetyl Cysteine Ethyl Ester. Subjects will report to the lab on three different occasions to consume the products, using a randomized cross-over design, and blood will be collected periodically (for the initial 8 hours and then again at 24 hours) per standard, routinely used pharmacokinetic /pharmacodynamic study protocols for evaluation of circulating glutathione concentrations. The hypothesis for this study is that the combination of N-Acetyl Cysteine Ethyl Ester + glycine will yield the greatest increase in glutathione, followed by N-Acetyl Cysteine Ethyl Ester, followed by N-Acetyl Cysteine. These findings will provide initial evidence specific to the bioavailability of these treatments following a single acute ingestion and may guide future recommendations regarding routine use.

DETAILED DESCRIPTION:
One method of enhancing the uptake of N-Acetyl Cysteine following oral ingestion is to use the ethyl ester form, referred to as N-Acetyl Cysteine Ethyl Ester, which exerts remarkable antioxidant potential . N-Acetyl Cysteine Ethyl Ester is also available as a dietary supplement, has been well-investigated and known to be much more effective than traditional N-Acetyl Cysteine, in terms of elevating glutathione levels. In addition, recent work indicates that inclusion of the amino acid glycine along with very high dose N-Acetyl Cysteine results in an increase in glutathione, which may have health enhancing benefits for a variety of conditions. Such an elevation in glutathione may provide for antioxidant benefits which can reduce oxidative stress and possibly aid various aspects of overall health, as oxidative stress is associated with disease and aging.

The study compares three different formulations containing N-Acetyl Cysteine, with regards to acute absorption over a 24-hour period, following single ingestion. The formulations are traditional N-Acetyl Cysteine, N-Acetyl Cysteine Ethyl Ester, and a product containing a combination of N-Acetyl Cysteine Ethyl Ester, glycine, and two minerals with antioxidant potential (selenium and molybdenum) that might enhance the effect of N-Acetyl Cysteine Ethyl Ester. Subjects will report to the lab on three different occasions to consume the products, using a randomized cross-over design, and blood will be collected periodically (for the initial 8 hours and then again at 24 hours) per standard, routinely used pharmacokinetic /pharmacodynamic study protocols for evaluation of circulating glutathione concentrations. The hypothesis for this study is that the combination of N-Acetyl Cysteine Ethyl Ester + glycine will yield the greatest increase in glutathione, followed by N-Acetyl Cysteine Ethyl Ester, followed by N-Acetyl Cysteine. These findings will provide initial evidence specific to the bioavailability of these treatments following a single acute ingestion and may guide future recommendations regarding routine use.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active (2 or more days per week of exercise for greater than 30 minutes/day)
* Body mass index between 18-29.9 kilograms per meter squared
* fast overnight (greater than 10 hours)
* willing to adhere to study procedures

Exclusion Criteria:

* tobacco user
* chronic disease, including diagnosed digestive disorders
* allergy or sensitivity to study product
* alcohol consumption within 24 hours of study visit
* caffeine consumption within 24 hours of study visit
* active infection or illness
* lactating, pregnant, planning to become pregnant during study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Area under the concentration curve for glutathione | 24 hour period following supplement ingestion
  The area under the concentration curve for reduced glutathione over oxidized glutathione will be calculated for each supplement.
Terminal Half-life of glutathione | 24 hour period following supplement ingestion
  The terminal half-life of reduced glutathione over oxidized glutathione will be calculated for each supplement
Peak concentration of glutathione | 24 hour period following supplement ingestion
  The peak concentration of reduced glutathione over oxidized glutathione will be determined for each supplement
Time to maximum concentration | 24 hour period following supplement ingestion
  The time to reaching the maximum concentration of reduced glutathione over oxidized glutathione will be determined for each supplement
Lag time | 24 hour period following supplement ingestion
  The lag time of each supplement will be determined.
Apparent volume distribution during terminal elimination phase | 24 hour period following supplement ingestion
  The apparent volume distribution during terminal elimination phase will be determined for reduced glutathione over oxidized glutathione
Oral Clearance of glutathione | 24 hour period following supplement ingestion
  The oral clearance of each supplement will be determined.

SECONDARY OUTCOMES:
Blood Malondialdehyde | 0 min prior to supplement ingestion (baseline)
  The concentration of malondialdehyde in blood will be measured in millimoles per liter
Blood Malondialdehyde | 2 hours following supplement ingestion
  The concentration of malondialdehyde in blood will be measured millimoles per liter
Blood Malondialdehyde | 4 hours following supplement ingestion
  The concentration of malondialdehyde in blood will be measured millimoles per liter
Blood Malondialdehyde | 8 hours following supplement ingestion
  The concentration of malondialdehyde in blood will be measured millimoles per liter
Blood Malondialdehyde | 24 hours following supplement ingestion
  The concentration of malondialdehyde in blood will be measured millimoles per liter
Blood Advanced Oxidation Protein Products | 0 min prior to supplement ingestion (baseline)
  The concentration of blood advanced oxidation protein products will be measured in units of micromoles Chloramine per liter
Blood Advanced Oxidation Protein Products | 2 hours following supplement ingestion
  The concentration of blood advanced oxidation protein products will be measured in units of micromoles Chloramine per liter
Blood Advanced Oxidation Protein Products | 4 hours following supplement ingestion
  The concentration of blood advanced oxidation protein products will be measured in units of micromoles Chloramine per liter
Blood Advanced Oxidation Protein Products | 8 hours following supplement ingestion
  The concentration of blood advanced oxidation protein products will be measured in units of micromoles Chloramine per liter
Blood Advanced Oxidation Protein Products | 24 hours following supplement ingestion
  The concentration of blood advanced oxidation protein products will be measured in units of micromoles Chloramine per liter
Brunel Mood Scale | 0 min prior to supplement ingestion (baseline)
  The brunel mood scale is a 24-item scale that consists of basic mood descriptors rated by the subject using a 5-point Likert scale where a score of 0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, and 4 = extremely.
Brunel Mood Scale | 2 hours following supplement ingestion
  The brunel mood scale is a 24-item scale that consists of basic mood descriptors rated by the subject using a 5-point Likert scale where a score of 0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, and 4 = extremely.
Brunel Mood Scale | 4 hours following supplement ingestion
  The brunel mood scale is a 24-item scale that consists of basic mood descriptors rated by the subject using a 5-point Likert scale where a score of 0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, and 4 = extremely.
Brunel Mood Scale | 8 hours following supplement ingestion
  The brunel mood scale is a 24-item scale that consists of basic mood descriptors rated by the subject using a 5-point Likert scale where a score of 0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, and 4 = extremely.
Brunel Mood Scale | 24 hours following supplement ingestion
  The brunel mood scale is a 24-item scale that consists of basic mood descriptors rated by the subject using a 5-point Likert scale where a score of 0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, and 4 = extremely.
Subjective Feelings | 0 min prior to supplement ingestion (baseline)
  Subjective feelings will be self-assessed by subjects for energy, mood, motivation, focus, attention, irritability, and jitters the subject using a 100 mm visual analog scale from 0 (none) to 10 (extreme)
Subjective Feelings | 2 hours following supplement ingestion
  Subjective feelings will be self-assessed by subjects for energy, mood, motivation, focus, attention, irritability, and jitters the subject using a 100 mm visual analog scale from 0 (none) to 10 (extreme)
Subjective Feelings | 4 hours following supplement ingestion
  Subjective feelings will be self-assessed by subjects for energy, mood, motivation, focus, attention, irritability, and jitters the subject using a 100 mm visual analog scale from 0 (none) to 10 (extreme)
Subjective Feelings | 8 hours following supplement ingestion
  Subjective feelings will be self-assessed by subjects for energy, mood, motivation, focus, attention, irritability, and jitters the subject using a 100 mm visual analog scale from 0 (none) to 10 (extreme)
Subjective Feelings | 24 hours following supplement ingestion
  Subjective feelings will be self-assessed by subjects for energy, mood, motivation, focus, attention, irritability, and jitters the subject using a 100 mm visual analog scale from 0 (none) to 10 (extreme)

OTHER OUTCOMES:
Heart Rate | 0 min prior to supplement ingestion (baseline)
  Heart Rate will be assessed in beats per minute using an automated blood pressure cuff.
Heart Rate | 0.25 hours following supplement ingestion
  Heart Rate will be assessed in beats per minute using an automated blood pressure cuff.
Heart Rate | 0.5 hours following supplement ingestion
  Heart Rate will be assessed in beats per minute using an automated blood pressure cuff.
Heart Rate | 1 hour following supplement ingestion
  Heart Rate will be assessed in beats per minute using an automated blood pressure cuff.
Heart Rate | 1.5 hours following supplement ingestion
  Heart Rate will be assessed in beats per minute using an automated blood pressure cuff.
Heart Rate | 2 hours following supplement ingestion
  Heart Rate will be assessed in beats per minute using an automated blood pressure cuff.
Heart Rate | 4 hours following supplement ingestion
  Heart Rate will be assessed in beats per minute using an automated blood pressure cuff.
Heart Rate | 6 hours following supplement ingestion
  Heart Rate will be assessed in beats per minute using an automated blood pressure cuff.
Heart Rate | 8 hours following supplement ingestion
  Heart Rate will be assessed in beats per minute using an automated blood pressure cuff.
Heart Rate | 24 hours following supplement ingestion
  Heart Rate will be assessed in beats per minute using an automated blood pressure cuff.
Diastolic Blood Pressure | 0 min prior to supplement ingestion (baseline)
  Diastolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Diastolic Blood Pressure | 0.25 hours following supplement ingestion
  Diastolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Diastolic Blood Pressure | 0.5 hours following supplement ingestion
  Diastolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Diastolic Blood Pressure | 1 hour following supplement ingestion
  Diastolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Diastolic Blood Pressure | 1.5 hours following supplement ingestion
  Diastolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Diastolic Blood Pressure | 2 hours following supplement ingestion
  Diastolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Diastolic Blood Pressure | 4 hours following supplement ingestion
  Diastolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Diastolic Blood Pressure | 6 hours following supplement ingestion
  Diastolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Diastolic Blood Pressure | 8 hours following supplement ingestion
  Diastolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Diastolic Blood Pressure | 24 hours following supplement ingestion
  Diastolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Systolic Blood Pressure | 0 min prior to supplement ingestion (baseline)
  Systolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Systolic Blood Pressure | 0.25 hours following supplement ingestion
  Systolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Systolic Blood Pressure | 0.5 hours following supplement ingestion
  Systolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Systolic Blood Pressure | 1 hour following supplement ingestion
  Systolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Systolic Blood Pressure | 1.5 hours following supplement ingestion
  Systolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Systolic Blood Pressure | 2 hours following supplement ingestion
  Systolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Systolic Blood Pressure | 4 hours following supplement ingestion
  Systolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Systolic Blood Pressure | 6 hours following supplement ingestion
  Systolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Systolic Blood Pressure | 8 hours following supplement ingestion
  Systolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.
Systolic Blood Pressure | 24 hours following supplement ingestion
  Systolic blood pressure will be assessed in millimeters mercury using an automated blood pressure cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States